CLINICAL TRIAL: NCT00572169
Title: A Phase II Study Incorporating Bone Marrow Microenvironment (ME) - Co-Targeting Bortezomib Into Tandem Melphalan-Based Autotransplants With DTPACE for Induction/Consolidation and Thalidomide + Dexamethasone for Maintenance
Brief Title: UARK 2006-66, Total Therapy 3B: An Extension of UARK 2003-33 Total Therapy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 72023
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Thalidomide; Dexamethasone; Calcium Dobesilate; Doxorubicin; Cisplatin; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VDTPACE (Experimental): Velcade, Dexamethasone, Thalidomide, Cisplatinin, Adriamycin, Cyclophosphamide and Etoposide
  Interventions: Drug: Velcade; Drug: Thalidomide; Drug: Dexamethasone; Drug: Adriamycin; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Etoposide

INTERVENTIONS:
Drug: Velcade — Will be given in central venous catheter
  Other Names: Bortezomib, PS-341
Drug: Thalidomide — Capsule taken by mouth
  Other Names: Thalomid
Drug: Dexamethasone — A pill taken by mouth
  Other Names: Decadron, NSC-34521
Drug: Adriamycin — Given into the vein (IV) by a continuous infusion through a central catheter
  Other Names: Doxorubicin, NSC-123127
Drug: Cisplatin — Given into the vein (IV) by a continuous infusion through a central catheter
  Other Names: Cis-diamminedichloroplatinum [CDDP], Platinol, NSC-119875
Drug: Cyclophosphamide — Given into the vein (IV) by a continuous infusion through a central catheter
  Other Names: Cytoxan, NSC-26271
Drug: Etoposide — Given into the vein (IV) by a continuous infusion through a central catheter
  Other Names: VP-16), Vepesid®, Ethylidene-Lignan P., NSC-141540

SUMMARY:
With this study - Total Therapy IIIB - researchers are extending the findings of Total Therapy III based what they have learned from the first two studies (Total Therapy I and II), with new research strategies designed to explore why chromosome abnormalities found in persons with multiple myeloma affect the outcome of drug therapy used in this disease."

DETAILED DESCRIPTION:
It is well known that myeloma patients with chromosome abnormalities are at higher risk because their disease tends to be more aggressive and does not respond to treatment as well as patients without chromosome abnormalities. When researchers at the Myeloma Institute looked at the results of Total Therapy II, they found that although research subjects with chromosome abnormalities had better outcomes (how many responded, and how long they survived) than those treated with standard chemotherapy; still their outcomes did not improve significantly with Total Therapy II, when compared to Total Therapy I.

The research in this new study is designed to target this high-risk group of individuals with chromosomal abnormalities. However, it is hoped that both groups of research participants - those with and without chromosome abnormalities - will derive benefit from changes made in this new research study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed active MM requiring treatment. Patients with a previous history of smoldering myeloma will be eligible if there is evidence of progressive disease requiring chemotherapy.
* Protein criteria must be present (quantifiable serum M-component of IgG, IgA, IgD, or IgE; urinary kappa or lambda light chain; or serum free light chain (SFLC) levels in order to evaluate response. Non-secretory patients are eligible provided the patient has > 20% plasmacytosis OR multiple (>3) focal plasmacytomas or focal lesions on MRI OR diffuse hyperintense signal on STIR images in the absence of hematopoietic growth factors.
* Patients must have received no more than one cycle or one month of prior chemotherapy for this disease. Patients may have received prior radiotherapy provided approval has been obtained by the Principal Investigator.
* Patients must be <75 years of age at the time of initial registration.
* Ejection fraction by ECHO or MUGA ≥ 40% performed within 60 days prior to registration.
* Patients must have adequate pulmonary function studies > 50% of predicted on mechanical aspects (FEV1, FVC, etc) and diffusion capacity (DLCO) > 50% of predicted, within 60 days of registration. If the patient is unable to complete pulmonary function tests due to MM related pain or condition, exception may be granted if the principal investigator documents that the patient is a candidate for high dose therapy.
* Patients must have a performance status of 0-2 based on SWOG criteria. Patients with a poor performance status (3-4), based solely on bone pain, will be eligible.
* All patients must be informed of the investigational nature of this study and must have signed an IRB-approved informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Platelet count < 30 x 109/L, unless myeloma-related.
* 5.1.2.2 Grade > 2 peripheral neuropathy.
* Hypersensitivity to bortezomib, boron, or mannitol.
* Uncontrolled diabetes.
* Recent (< 6 months) myocardial infarction, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension, or difficult to control cardiac arrhythmias.
* Evidence of chronic obstructive or chronic restrictive pulmonary disease.
* Patients must not have light chain deposition disease or creatinine > 3 mg/dl
* Patients must not have prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has not received treatment for one year prior to enrollment. Other cancers will only be acceptable if the patient's life expectancy exceeds five years.
* Patients must not have significant co-morbid medical conditions or uncontrolled life threatening infection.
* Pregnant or nursing women. Women of child-bearing potential must have a negative pregnancy test documented within one week of registration. Women and men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2006-11; Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
To find out if outcomes of participants in this study will be better when compared to individuals who participated in Total Therapy II, especially those with chromosome abnormalities. | 48 months

SECONDARY OUTCOMES:
To find out if outcomes and incidence of toxicities of participants in this study will be better when compared to individuals who participated in Total Therapy III. | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Morgan, MD, PhD, Principal Investigator — UAMS Myeloma Institute for Research and Therapy
Locations (1):
- University of Arkansas for Medical Sciences/Myeloma Institute, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Al Hadidi S, Ababneh OE, Schinke CD, Thanendrarajan S, Bailey C, Smith R, Panozzo S, Alapat D, Cottler-Fox M, Tricot G, Shaughnessy JD Jr, Zhan F, Sawyer J, Barlogie B, Zangari M, van Rhee F. Three years of maintenance with VRD in multiple myeloma: results of total therapy IIIB with a 15-year follow-up. Blood Adv. 2024 Feb 13;8(3):703-707. doi: 10.1182/bloodadvances.2023011601. PMID 38052037
- [Derived] Pawlyn C. High-risk myeloma: a challenge to define and to determine the optimal treatment. Lancet Haematol. 2021 Jan;8(1):e4-e6. doi: 10.1016/S2352-3026(20)30361-6. Epub 2020 Dec 22. No abstract available. PMID 33357481
- [Derived] Usmani SZ, Sawyer J, Rosenthal A, Cottler-Fox M, Epstein J, Yaccoby S, Sexton R, Hoering A, Singh Z, Heuck CJ, Waheed S, Chauhan N, Johann D, Abdallah AO, Muzaffar J, Petty N, Bailey C, Crowley J, van Rhee F, Barlogie B. Risk factors for MDS and acute leukemia following total therapy 2 and 3 for multiple myeloma. Blood. 2013 Jun 6;121(23):4753-7. doi: 10.1182/blood-2012-11-466961. Epub 2013 Apr 19. PMID 23603914
- [Derived] Usmani SZ, Mitchell A, Waheed S, Crowley J, Hoering A, Petty N, Brown T, Bartel T, Anaissie E, van Rhee F, Barlogie B. Prognostic implications of serial 18-fluoro-deoxyglucose emission tomography in multiple myeloma treated with total therapy 3. Blood. 2013 Mar 7;121(10):1819-23. doi: 10.1182/blood-2012-08-451690. Epub 2013 Jan 10. PMID 23305732
- [Derived] Usmani SZ, Heuck C, Mitchell A, Szymonifka J, Nair B, Hoering A, Alsayed Y, Waheed S, Haider S, Restrepo A, Van Rhee F, Crowley J, Barlogie B. Extramedullary disease portends poor prognosis in multiple myeloma and is over-represented in high-risk disease even in the era of novel agents. Haematologica. 2012 Nov;97(11):1761-7. doi: 10.3324/haematol.2012.065698. Epub 2012 Jun 11. PMID 22689675
- [Derived] Usmani SZ, Sexton R, Hoering A, Heuck CJ, Nair B, Waheed S, Al Sayed Y, Chauhan N, Ahmad N, Atrash S, Petty N, van Rhee F, Crowley J, Barlogie B. Second malignancies in total therapy 2 and 3 for newly diagnosed multiple myeloma: influence of thalidomide and lenalidomide during maintenance. Blood. 2012 Aug 23;120(8):1597-600. doi: 10.1182/blood-2012-04-421883. Epub 2012 Jun 6. PMID 22674807